CLINICAL TRIAL: NCT04596332
Title: Central Venous Pressure Monitoring is Associated With Improved Prognosis of High-risk Operating Patients During Perioperative Period
Brief Title: Central Venous Pressure Monitoring and Prognosis of High-risk Operating Patients
Status: Completed | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Xiuling Shang, Department of Critical Care Medicine, Fujian Provincial Hospital, Fujian Provincial Hospital
Other Study IDs: K2018-09-006
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Central Venous Pressure
Keywords: perioperative; central venous pressure; fluid management; acute renal injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Patients with the initial central venous pressure(CVP1) <8 mm Hg
  Interventions: Other: no intervention measures
- Group B: Patients with 8≤CVP1≤12mm Hg
  Interventions: Other: no intervention measures
- Group C: Patients with CVP1>12 mm Hg
  Interventions: Other: no intervention measures

INTERVENTIONS:
Other: no intervention measures — Because this study was a retrospective study, no intervention measures were implemented for the patients enrolled.

SUMMARY:
While central venous pressure measurement is used to guide fluid management in high risk surgical patients during perioperative period, the relationship between the value of central venous pressure and organ dysfunction and prognosis of high-risk operating patients is unknow. In this study, we conducted a retrospective study of the relationship between the initial levels of CVP with organ dysfunction, the severity of illness, the length of ICU stay, and prognosis of critically ill patients.

DETAILED DESCRIPTION:
Although less than 15% of high-risk patients (elderly or with limited cardiopulmonary reserves) undergo surgery, these patients account for 80% of hospital deaths. The requirements for hemodynamic monitoring to critical patients during perioperative period reach are of maximal importance, for two major reasons: (i) absolute or relative volume deficiency often occurs in postoperative patients due to preoperative fasting, intraoperative bleeding and non-dominant fluid loss caused by vasodilation and fluid redistribution caused by anesthesia; (ii) insufficient fluid replacement may lead to increased postoperative organ complications and poor wound healing. Adequate and goal-oriented hemodynamic monitoring combined with early and appropriate treatment can improve the prognosis of high-risk surgical patients.

Central venous pressure is a localized parameter of the superior vena cava or the right atrium and is closely related to the right ventricular end-diastolic pressure. With volume overload, CVP levels may be abnormally elevated. Maintaining central venous pressure as low as possible is conducive to the recovery of internal organs during haemodynamic treatment, especially for the kidney, intestine, and brain, etc. However, elevated central venous pressure (CVP) occurs frequently in critical care settings, including postoperative critical patients. In this study, we conducted a retrospective study of the relationship between the initial levels of CVP with organ dysfunction, the severity of illness, the length of ICU stay, and prognosis of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.⑵ All patients undergoing surgery and admitted to our intensive care unit (ICU) directly after surgery were enrolled into the respective study.⑶ They stayed in the ICU more than 48 hours with central venous pressure monitored for more than 48 hours.

Exclusion Criteria:

* Patients who were in pregnancy. ⑵Older than 80 years. ⑶Underwent cardiac surgery or had chronic kidney disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-center, retrospective, observational study enrolled 196 patients undergoing high-risk surgery who admitted to surgical intensive care unit(SICU) directly after operation from Feb 1,2014 to Mar 31,2018.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 28-day
  28-day mortality, length of stay in intensive care unit and hospitalization, surgical complications

SECONDARY OUTCOMES:
Secondary Outcome | 1-day
  Comparison of perioperative fluid management in each group

CONTACTS AND LOCATIONS:
Overall Officials: Jiafang Wu, M.D., Principal Investigator — Department of Critical Care Medicine, Fujian Provincial Hospital

IPD SHARING:
Plan to Share IPD: No